CLINICAL TRIAL: NCT03109600
Title: A Randomized, Observer Blinded, Comparative, Phase I Safety Study in Two Age De-escalating Cohorts to Assess the Safety and Immunogenicity of Vi-DT Typhoid Conjugate Vaccine (Bio Farma) in Adults and Children (Phase I)
Brief Title: Safety and Immunogenicity of Vi-DT Typhoid Conjugate Vaccine (Bio Farma) in Adults and Children (Phase I)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PT Bio Farma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Typhoid 0116
Record Dates: First submitted 2016-11-01; First posted 2017-04-12 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2017-07

CONDITIONS: Safety Issues
MeSH Terms: interventions — Vi polysaccharide vaccine, typhoid; Pneumococcal Vaccines

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Vi-DT (Bio Farma) (Experimental): 2 dose of 0.5 ml of Vi-DT Conjugated typhoid vaccine
  Interventions: Biological: Vi-DT (Bio Farma)
- Vi polysaccharide vaccine (Active Comparator): 1 dose of 0.5 ml Vi polysaccharide vaccine + 1 dose of Influenzae Vaccine
  Interventions: Biological: Vi polysaccharide vaccine; Biological: Influenzae vaccine
- Vi-DT (Bio Farma) ~ Children (Experimental): 2 dose of 0.5 ml of Vi-DT Conjugated typhoid vaccine
  Interventions: Biological: Vi-DT (Bio Farma)
- Vi polysaccharide vaccine ~ Children (Active Comparator): 1 dose of 0.5 ml Vi polysaccharide vaccine + 1 dose of Pneumococcal Conjugate Vaccine
  Interventions: Biological: Vi polysaccharide vaccine; Biological: Pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: Vi-DT (Bio Farma) — Typhoid Conjugate Vaccine
  Arms: Vi-DT (Bio Farma); Vi-DT (Bio Farma) ~ Children
Biological: Vi polysaccharide vaccine — Vi polysaccharide vaccine
  Arms: Vi polysaccharide vaccine; Vi polysaccharide vaccine ~ Children
Biological: Influenzae vaccine — 1 dose of Influenzae vaccine
  Arms: Vi polysaccharide vaccine
Biological: Pneumococcal conjugate vaccine — 1 dose of Pneumococcal conjugate Vaccine
  Arms: Vi polysaccharide vaccine ~ Children

SUMMARY:
This study is to assess the safety of Vi-DT vaccine in adults and children.

DETAILED DESCRIPTION:
To describe the safety of this vaccine following first and second dose immunization.

To assess preliminary information of immunogenicity following Vi-DT vaccine immunization.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy
2. Subjects/Parents have been informed properly regarding the study and signed the informed consent form
3. Subject/Parents will commit to comply with the instructions of the investigator and the schedule of the trial

Exclusion Criteria:

1. Subject concomitantly enrolled or scheduled to be enrolled in another trial
2. Evolving mild, moderate or severe illness, especially infectious diseases or fever (axillary temperature ³ 37.5°C )
3. Known history of allergy to any component of the vaccines
4. History of uncontrolled coagulopathy or blood disorders contraindicating intramuscular injection
5. Subject who has received in the previous 4 weeks a treatment likely to alter the immune response (intravenous immunoglobulins, blood-derived products or long term corticotherapy (> 2 weeks).
6. Any abnormality or chronic disease which according to the investigator might interfere with the assessment of the trial objectives
7. Pregnancy & lactation (Adults)
8. Individuals who have previously received any vaccines against typhoid fever.
9. Subjects already immunized with any vaccine within 4 weeks prior and expect to receive other vaccines within 60 days following the first dose.
10. Individuals who have a previously ascertained typhoid fever.
11. History of alcohol or substance abuse.
12. Subject planning to move from the study area before the end of study period.

Ages: 2 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2017-09-28 (Actual); Study Completion 2018-02-19 (Actual)

PRIMARY OUTCOMES:
Local reaction and systemic event after vaccination | 28 days
  Percentage of subjects with at least one immediate reaction (local reaction or systemic event) after vaccination.

SECONDARY OUTCOMES:
Adverse events after vaccination | 28 days
  Percentage of subjects with at least one of these adverse events, solicited or not, within 24 h, 48h, 72h and 28 days after each vaccination.
Serious adverse events after vaccination | 28 days
  Number and percentage of subjects with serious adverse event from inclusion until 28 day after vaccination and up to 6 months after the last vaccination.
Routine laboratory evaluation that probably related to the vaccination. | 7 days
  Deviation from routine blood laboratory, kidney and liver function laboratory evaluation that probably related to the vaccination.
Preliminary assessment of immunogenicity of typhoid conjugated vaccine (Vi-DT) | 28 days
  Percentage of subjects with > 4 times increasing antibody
Geometric Mean Titers (GMT) following immunization | 28 days
  Geometric Mean Titers (GMT) 28 days following immunization

CONTACTS AND LOCATIONS:
Overall Officials: Bernie Endyarni, MD, Principal Investigator — Faculty of Medicine, University of Indonesia
Locations (2):
- Indonesia (2):
  - Puskesmas Jatinegara, Jakarta, DKI Jaya
  - Jatinegara Primary Health Center, Jakarta

IPD SHARING:
Plan to Share IPD: No